CLINICAL TRIAL: NCT00667251
Title: A Randomized, Open-Label, Phase III Study of Taxane Based Chemotherapy With Lapatinib or Trastuzumab as First-Line Therapy for Women With HER2/Neu Positive Metastatic Breast Cancer
Brief Title: Chemotherapy and Lapatinib or Trastuzumab in Treating Women With HER2/Neu-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108919; CLAP016A2303 (Other: Novartis); CAN-NCIC-MA31 (Other Grant/Funding Number: NCI US - Physician Data Query); 2007-004568-27 (EudraCT Number); CDR0000594764 (Other: PDQ); EGF108919 (Other: GSK)
Record Dates: First submitted 2008-04-25; First posted 2008-04-28 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; HER2-positive breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel; Lapatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lapatinib (Active Comparator): Plus taxane based chemotherapy
  Interventions: Drug: docetaxel; Drug: lapatinib ditosylate; Drug: paclitaxel
- Trastuzumab (Active Comparator): Plus taxane based chemotherapy.
  Interventions: Biological: trastuzumab; Drug: docetaxel; Drug: paclitaxel

INTERVENTIONS:
Biological: trastuzumab — IV q weekly (loading dose 4mg/kg; subsequent doses 2mg/kg) or IV q 3 weekly (loading dose 8mg/kg, subsequent doses 6mg/kg).
  Arms: Trastuzumab
Drug: docetaxel — 75mg/m2 IV q 3 weekly, day 1 of a 3 week cycle for 8 cycles plus G-CSF (when given together with lapatinib).
Drug: lapatinib ditosylate — 1250 mg once daily (while given with taxane). 1500mg once daily (when given alone after taxane completion).
  Arms: Lapatinib
Drug: paclitaxel — 80mg/m2 IV q weekly days 1, 8 and 15 of a 4-week cycle for 6 cycles.

SUMMARY:
This was a multi-center, multinational, randomized, open-label, Phase III study comparing combination taxane-based chemotherapy plus lapatinib to combination taxane-based chemotherapy plus trastuzumab in women with documented evidence of human epidermal growth factor receptor 2 (HER2) positive metastatic breast cancer (MBC) (by local or central laboratory testing) who had received no prior chemotherapy or HER2 targeted therapy in the metastatic setting.

DETAILED DESCRIPTION:
Subjects were stratified by

* Prior (neo) adjuvant HER2/neu targeted therapy (yes, no)
* Prior (neo) adjuvant taxane chemotherapy (yes, no)
* Planned taxane treatment (once weekly paclitaxel versus docetaxel once every 3 weeks)
* Liver metastasis (yes, no)

Subjects were randomized 1:1 to the following treatments to a planned sample size of approximately 600 subjects (to achieve 536 centrally confirmed HER2 positive subjects):

* Taxane based chemotherapy plus lapatinib for 24 weeks followed by single agent lapatinib
* Taxane based chemotherapy plus trastuzumab for 24 weeks followed by single agent trastuzumab

The choice of taxane (once weekly paclitaxel versus docetaxel once every 3 weeks) was at the discretion of the treating physician and was specified at the time of subject randomization.

A protocol-specified interim analysis was conducted on 27-Apr-2012, following which the participants in the Lapatinib plus taxane based chemotherapy arm could cross over to Taxane based chemotherapy plus Trastuzumab.

ELIGIBILITY:
Key inclusion criteria:

* Histologically confirmed adenocarcinoma of the breast.
* MBC (stage IV) at primary diagnosis or at relapse after curative intent therapy.
* Local or central laboratory confirmed HER2/neu overexpressing and/or amplified disease in the invasive component of the primary or metastatic lesion as defined by:

  1. 3+ over expression by immunohistochemistry (IHC) (>30% of invasive tumour cells);
  2. 2+ or 3+ (in 30% or less neoplastic cells) overexpression by IHC analysis AND fluorescence or chromogenic in situ hybridization (FISH/CISH) test demonstrating HER2/neu gene amplification;
  3. HER2/neu gene amplification by FISH/CISH [>6 HER2/neu gene copies per nucleus, or a FISH/CISH ratio (HER2 gene copies to chromosome 17 signals) of >=2.2]
* Subjects must have had evidence of metastatic disease, but measurable disease was not mandatory. To be considered evaluable for overall response rate (CR and PR), subjects must have had at least 1 measurable lesion as follows:

  1. X-ray, physical exam >=20 mm.
  2. Conventional computed tomography (CT) scan, magnetic resonance imaging (MRI) >=20 mm.
  3. Spiral CT scan >=10 mm.

Key exclusion criteria:

* Subjects with a history of other malignancies, except: adequately treated ductal carcinoma in-situ or lobular carcinoma in-situ, adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumor (non-breast) curatively treated with no evidence of disease for >=5 years.
* Subjects who had received prior chemotherapy, immunotherapy, biologic therapy or HER2/neu targeted therapy for recurrent or MBC.
* Subjects receiving ongoing anti-cancer treatment or other investigational anti-cancer agents for breast cancer or subjects who had used an investigational drug within 30 days or 5 half-lives (if known), whichever was longer, preceding the date of randomization.
* Subjects with: CNS metastases (including leptomeningeal involvement), serious cardiac illness, peripheral neuropathy grade 2 or greater, subjects with gastrointestinal tract disease, subjects receiving CYP3A4 inhibitors or inducers, and subjects with history of allergic or hypersensitivity reactions to any study drug or their excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2008-10-07 (Actual); Primary Completion 2012-08-01 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (237):
- United States (52):
  - Novartis Investigative Site, Anchorage, Alaska
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Berkeley, California
  - Novartis Investigative Site, Highland, California
  - Novartis Investigative Site, Montebello, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Greenwich, Connecticut
  - Novartis Investigative Site, Southington, Connecticut
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigative Site, Trumbull, Connecticut
  - Novartis Investigative Site, Waterbury, Connecticut
  - Novartis Investigative Site, Kissimmee, Florida
  - Novartis Investigative Site, Loxahatchee Groves, Florida
  - Novartis Investigative Site, New Port Richey, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Lawrenceville, Georgia
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, Post Falls, Idaho
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Oak Lawn, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Goshen, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Munster, Indiana
  - Novartis Investigative Site, New Albany, Indiana
  - Novartis Investigative Site, Towson, Maryland
  - Novartis Investigative Site, Wheaton, Maryland
  - Novartis Investigative Site, Bozeman, Montana
  - Novartis Investigative Site, Grand Island, Nebraska
  - Novartis Investigative Site, Kearney, Nebraska
  - Novartis Investigative Site, Denville, New Jersey
  - Novartis Investigative Site, Parsippany, New Jersey
  - Novartis Investigative Site, Cooperstown, New York
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Wooster, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Chesapeake, Virginia
  - Novartis Investigative Site, Salem, Virginia
  - Novartis Investigative Site, Bellevue, Washington
  - Novartis Investigative Site, Kirkland, Washington
  - Novartis Investigative Site, Mount Vernon, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Sequim, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Wenatchee, Washington
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (8):
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Cipolletti, Río Negro Province
  - Novartis Investigative Site, Viedma, Río Negro Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán
  - Novartis Investigative Site, Santa Fe
- Australia (13):
  - Novartis Investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Tweed Heads, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Kurralta Park, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Wodonga, Victoria
  - Novartis Investigative Site, Subiaco, Western Australia
- Belgium (4):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Namur
- Canada (23):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Kelowna, British Columbia
  - Novartis Investigative Site, Surrey, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Saint John, New Brunswick
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Sault Ste. Marie, Ontario
  - Novartis Investigative Site, St. Catharines, Ontario
  - Novartis Investigative Site, Thunder Bay, Ontario
  - Novartis Investigative Site, Charlottetown, Prince Edward Island
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Regina, Saskatchewan
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- France (8):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Metz-Tessy
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
- Germany (32):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Coburg, Bavaria
  - Novartis Investigative Site, Eggenfelden, Bavaria
  - Novartis Investigative Site, Fürth, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Rosenheim, Bavaria
  - Novartis Investigative Site, Weiden, Bavaria
  - Novartis Investigative Site, Fürstenwalde, Brandenburg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Fulda, Hesse
  - Novartis Investigative Site, Lich, Hesse
  - Novartis Investigative Site, Goslar, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Leer, Lower Saxony
  - Novartis Investigative Site, Bielefeld, North Rhine-Westphalia
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Coesfeld, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Porta Westfalica, North Rhine-Westphalia
  - Novartis Investigative Site, Troisdorf, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Witten, North Rhine-Westphalia
  - Novartis Investigative Site, Koblenz, Rhineland-Palatinate
  - Novartis Investigative Site, Saarbrücken, Saarland
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Brandenburg
  - Novartis Investigative Site, Hamburg
- India (3):
  - Novartis Investigative Site, Bangalore
  - Novartis Investigative Site, Nagpur
  - Novartis Investigative Site, Pune
- Israel (5):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Holon
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Poria – Neve Oved
  - Novartis Investigative Site, Ramat Gan
- Italy (8):
  - Novartis Investigative Site, Lecce, Apulia
  - Novartis Investigative Site, Aviano (PN), Friuli Venezia Giulia
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Sora (FR), Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Sassari, Sardinia
  - Novartis Investigative Site, Prato (PO), Tuscany
  - Novartis Investigative Site, Chieti
- Japan (9):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Ehime
  - Novartis Investigative Site, Kagoshima
  - Novartis Investigative Site, Kanagawa
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Shizuoka
  - Novartis Investigative Site, Tokyo
- Mexico (3):
  - Novartis Investigative Site, Cuernavaca, Morelos
  - Novartis Investigative Site, Ciudad Obregón, Sonora
  - Novartis Investigative Site, Mexico City
- Netherlands (4):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Dordrecht
  - Novartis Investigative Site, Maastricht
- Poland (6):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Płock
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- Russia (10):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Lipetsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Ufa
- South Korea (3):
  - Novartis Investigative Site, Gyeonggi-do
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Songpa-gu, Seoul
- Spain (14):
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Alcorcón
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Badalona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Elche
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Jaén
  - Novartis Investigative Site, Lugo
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Majadahonda (Madrid)
  - Novartis Investigative Site, Pozuelo de Alarcon (Madrid)
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Taiwan (4):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan County
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Ukraine (4):
  - Novartis Investigative Site, Dnipro
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Sumy
- United Kingdom (22):
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Brighton
  - Novartis Investigative Site, Chelmsford
  - Novartis Investigative Site, Cheltenham
  - Novartis Investigative Site, Colchester
  - Novartis Investigative Site, Cottingham, Hull
  - Novartis Investigative Site, Derby
  - Novartis Investigative Site, Edmonton
  - Novartis Investigative Site, Guildford
  - Novartis Investigative Site, Harrogate
  - Novartis Investigative Site, Huddersfield
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Poole, Dorset
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Shrewsbury
  - Novartis Investigative Site, Sutton
  - Novartis Investigative Site, Whitchurch, Cardiff
  - Novartis Investigative Site, York

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Result] Gelmon KA, Boyle FM, Kaufman B, Huntsman DG, Manikhas A, Di Leo A, Martin M, Schwartzberg LS, Lemieux J, Aparicio S, Shepherd LE, Dent S, Ellard SL, Tonkin K, Pritchard KI, Whelan TJ, Nomikos D, Nusch A, Coleman RE, Mukai H, Tjulandin S, Khasanov R, Rizel S, Connor AP, Santillana SL, Chapman JA, Parulekar WR. Lapatinib or Trastuzumab Plus Taxane Therapy for Human Epidermal Growth Factor Receptor 2-Positive Advanced Breast Cancer: Final Results of NCIC CTG MA.31. J Clin Oncol. 2015 May 10;33(14):1574-83. doi: 10.1200/JCO.2014.56.9590. Epub 2015 Mar 16. PMID 25779558
- [Result] Ho D, Huang J, Chapman JW, Leitzel K, Ali SM, Shepherd L, Parulekar WR, Ellis CE, Crescnzo RJ, Zhu L, Virk S, Nomikos D, Aparicio S, Gelmon KA, Carney WP, Lipton A. Impact of serum HER2, TIMP-1, and CAIX on outcome for HER2+ metastatic breast cancer patients: CCTG MA.31 (lapatinib vs. trastuzumab). Breast Cancer Res Treat. 2017 Aug;164(3):571-580. doi: 10.1007/s10549-017-4273-x. Epub 2017 May 8. PMID 28484925
- [Result] Liu S, Chen B, Burugu S, Leung S, Gao D, Virk S, Kos Z, Parulekar WR, Shepherd L, Gelmon KA, Nielsen TO. Role of Cytotoxic Tumor-Infiltrating Lymphocytes in Predicting Outcomes in Metastatic HER2-Positive Breast Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2017 Nov 9;3(11):e172085. doi: 10.1001/jamaoncol.2017.2085. Epub 2017 Nov 9. PMID 28750133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 167 centers in 21 countries: Argentina (7), Australia (9), Belgium (3), Canada (19), France (5), Germany (23), India (3), Israel (4), Italy (7), Japan (12), Republic of Korea (4), Mexico (3), Netherlands (4), Poland (5), Russian Federation (7), Spain (14), Taiwan (4), Thailand (2), Ukraine (3), United Kingdom (18), United States (11).
Groups:
- Lapatinib (LTax/L): Lapatinib 1250 mg once daily. Taxane based chemotherapy: Paclitaxel 80 mg/m2 IV once weekly (Days 1, 8, and 15 of a 4-week cycle) OR Docetaxel 75 mg/m2 IV once every 3 weeks (Day 1 of a 3-week cycle) plus G-CSF: according to institutional standards. Followed by Lapatinib 1500 mg once daily until disease progression.
- Trastuzumab (TTax/T): Trastuzumab IV once weekly (loading dose 4 mg/kg, subsequent doses 2 mg/kg) and Paclitaxel 80 mg/m2 IV once weekly (Days 1, 8, and 15 of a 4-week cycle) OR Trastuzumab IV once every 3 weeks (loading dose 8 mg/kg, subsequent doses 6 mg/kg) and Docetaxel 75 mg/m2 IV once every 3 weeks (Day 1 of a 3-week cycle). Followed by Trastuzumab 6 mg/kg IV once every 3 weeks until disease progression.
Period: Overall Study
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Started (All randomized subjects were included in the Intent-to-Treat (ITT) population) | 326 | 326
Randomized Not Treated | 4 | 1
Crossed Over to Ttax/T After IA Results | 5 | 0
Central HER2 Positive (Subset of IIT population with centrally-confirmed human epidermal growth factor receptor 2 (HER2) positive tumors.) | 270 | 267
Safety Population (All randomized subjects who receive at least one dose of investigational product) | 322 | 325
Completed | 0 | 0
Not Completed | 326 | 326
Not completed — Disease progression | 232 | 203
Not completed — Toxicity | 44 | 23
Not completed — Subject Reached Protocol-Defined Stopping Criteria | 18 | 70
Not completed — Refused further treatment (not due to toxicity) | 8 | 7
Not completed — Symptomatic progression | 8 | 4
Not completed — Death | 6 | 11
Not completed — Intercurrent illness | 5 | 6
Not completed — Primary reason for withdrawal = missing | 1 | 1
Not completed — Randomized not Treated | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T) | Total
Number analyzed (Participants) | 326 | 326 | 652
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 260 | 263 | 523
  >=65 years | 66 | 63 | 129
Age, Continuous [Median (Full Range); unit: years] | 55.4 (26.6-87.1) [26.6 to 87.1] | 54.4 (29.3-84.3) [29.3 to 84.3] | 54.9 [26.6 to 87.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 326 | 326 | 652
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 34 | 68
  Not Hispanic or Latino | 288 | 283 | 571
  Unknown or Not Reported | 4 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 67 | 74 | 141
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 8 | 13
  White | 246 | 234 | 480
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: Participants]
  United States | 10 | 13 | 23
  Taiwan | 11 | 11 | 22
  Thailand | 9 | 12 | 21
  Spain | 19 | 19 | 38
  Ukraine | 4 | 4 | 8
  Russian Federation | 55 | 46 | 101
  Israel | 16 | 15 | 31
  United Kingdom | 33 | 32 | 65
  Italy | 5 | 8 | 13
  India | 4 | 4 | 8
  France | 5 | 5 | 10
  Mexico | 3 | 6 | 9
  Canada | 39 | 36 | 75
  Argentina | 8 | 4 | 12
  Poland | 7 | 12 | 19
  Belgium | 3 | 6 | 9
  Australia | 17 | 13 | 30
  Netherlands | 7 | 7 | 14
  Germany | 32 | 34 | 66
  Japan | 22 | 20 | 42
  Korea, Republic of | 17 | 19 | 36
Number of Participants with the Indicated Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status classifies participants according to their functional impairment, and scores indicate: 0, fully active; 1, ambulatory, restricted strenuous activity; 2, ambulatory, no work activity; 3, partially confined to bed; 4, totally confined in bed; 5, death.
  Participants
    0, fully active | 196 | 204 | 400
    1, ambulatory, restricted strenuous activity | 118 | 112 | 230
    2, ambulatory, no work activity | 12 | 10 | 22
Disease Status [Count of Participants; unit: Participants]
  Primary diagnosis | 138 | 138 | 276
  Progression after therapy | 187 | 187 | 374
  Missing | 1 | 1 | 2
Central review human epidermal growth factor receptor 2 (HER2) status [Count of Participants; unit: Participants]
  Positive Immunohistochemistry (IHC) or Fluorescence in situ hybridization (FISH) | 270 | 267 | 537
  Equivocal Immunohistochemistry (IHC) and Fluorescence in situ hybridization (FISH) | 9 | 5 | 14
  Negative Immunohistochemistry (IHC) and Fluorescence in situ hybridization (FISH) | 36 | 46 | 82
  Unknown | 11 | 8 | 19
Central review estrogen receptor (ER) status [Count of Participants; unit: Participants]
  Positive (>0) | 213 | 208 | 421
  Negative | 96 | 107 | 203
  Missing | 17 | 11 | 28
Central review progesterone receptor (PgR) status [Count of Participants; unit: Participants]
  Positive (>0) | 116 | 104 | 220
  Negative | 190 | 204 | 394
  Missing | 20 | 18 | 38
Central Review of Antigen KI-67 (ki67) [Geometric Mean (Full Range); unit: % cells positive] | 33.33 [0 to 100] | 31.43 [0 to 90] | 32.37 [0 to 100]
Central Review of Cytokeratin 5 (CK5) Status [Count of Participants; unit: Participants]
  Positive (>0) | 58 | 41 | 99
  Negative | 210 | 218 | 428
  Missing | 58 | 67 | 125
Central Review of epidermal growth factor receptor (EGFR) Status [Count of Participants; unit: Participants]
  Positive (>0) | 71 | 77 | 148
  Negative | 194 | 181 | 375
  Missing | 61 | 68 | 129
Prior (neo)adjuvant HER2 targeted therapy [Count of Participants; unit: Participants]
  Yes | 59 | 59 | 118
  No | 267 | 267 | 534
Prior (neo)adjuvant taxane chemotherapy [Count of Participants; unit: Participants]
  Yes | 65 | 69 | 134
  No | 261 | 257 | 518
Planned taxane treatment [Count of Participants; unit: Participants]
  Weekly paclitaxel | 146 | 146 | 292
  3-weekly docetaxel | 180 | 180 | 360
Liver metastasis [Count of Participants; unit: Participants]
  Yes | 149 | 150 | 299
  No | 177 | 176 | 353
Prior neoadjuvant therapy/Other chemotherapy [Count of Participants; unit: Participants]
  Yes | 146 | 161 | 307
  No | 180 | 165 | 345
Prior neoadjuvant therapy/Anthracyclines [Count of Participants; unit: Participants]
  Yes | 128 | 140 | 268
  No | 198 | 186 | 384
Prior neoadjuvant therapy/Other therapy [Count of Participants; unit: Participants]
  Yes | 5 | 2 | 7
  No | 321 | 323 | 644
  Missing | 0 | 1 | 1
Prior neoadjuvant/Metastatic radiotherapy [Count of Participants; unit: Participants]
  Yes | 138 | 149 | 287
  No | 187 | 176 | 363
  Missing | 1 | 1 | 2
Prior neoadjuvant/Metastatic endocrine therapy [Count of Participants; unit: Participants]
  Yes | 122 | 127 | 249
  No | 204 | 198 | 402
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) at the Time of Primary Results
Description: Progression-free survival (PFS) is the time from randomization to the earliest date of RECIST 1.0 assessment of disease progression (with radiological evidence), death from any cause, or censoring. Disease progression was assessed by the Investigator and defined by RECIST v1.0 as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of randomization until date of progression or date of death from any cause, whichever comes first, assessed up to approximately 39 months
Population: Intent-to-Treat (ITT) and centrally-confirmed HER2 positive populations
Measure: Median (Full Range); unit: Months
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 326 | 326
Months
  Intent-to-Treat (ITT) population | 8.97 [0.30 to 32.69] | 11.30 [0.30 to 38.54]
  centrally-confirmed HER2 positive population: number analyzed (Participants) | 270 | 267
  centrally-confirmed HER2 positive population | 9.13 [0.30 to 32.69] | 13.63 [0.30 to 38.54]
Statistical Analysis 1: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); PFS at the time of Primary Analysis (IIT population); Test type: Other; p = 0.0010, Log Rank; Hazard Ratio (HR) = 1.367, 95% CI 2-sided [1.133 to 1.648]
Statistical Analysis 2: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); PFS at the time of Primary Analysis (Central HER2+ population); Test type: Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 1.484, 95% CI 2-sided [1.204 to 1.829]

2. Secondary Outcome: Progression Free Survival (PFS) at the Time of Final Analysis
Description: Progression-free survival (PFS) is the time from randomization to the earliest date of RECIST 1.0 assessment of disease progression (with radiological evidence), death from any cause, or censoring. Disease progression was assessed by the Investigator and defined by RECIST v1.0 as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions. Subjects who crossover the treatment to Trastuzumab (TTax/T) after interim analysis, were censored at the last PFS assessment before crossover.
Time Frame: From date of randomization until date of progression or date of death from any cause, whichever comes first, assessed up to approximately 45 months
Population: Intent-to-Treat (ITT) and centrally-confirmed HER2 positive populations
Measure: Median (Full Range); unit: Months
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 326 | 326
Months
  Intent-to-Treat (ITT) population | 9.1 [8.5 to 10.8] | 11.5 [10.9 to 13.8]
  centrally-confirmed HER2 positive population: number analyzed (Participants) | 270 | 267
  centrally-confirmed HER2 positive population | 9.4 [8.5 to 11.0] | 13.8 [11.2 to 14.2]
Statistical Analysis 1: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); PFS at the time of Final Analysis (IIT population); Test type: Other; Hazard Ratio (HR) = 1.3722, 95% CI 2-sided [1.1466 to 1.6422] — Stratified HR for LTax/L versus TTax/T
Statistical Analysis 2: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); PFS at the time of Final Analysis (Central HER2+ population); Test type: Other; Hazard Ratio (HR) = 1.4968, 95% CI 2-sided [1.2251 to 1.8288] — Stratified HR for LTax/L versus TTax/T

3. Secondary Outcome: Overall Survival (OS) (IIT Population)
Description: Overall Survival (OS) was defined as the time interval between the date of randomization and the date of death from any cause. Subjects who were still alive at the time of the final analysis or became lost to follow-up, were censored at their last contact date. Subjects who crossover the treatment to Trastuzumab (TTax/T) after interim analysis, were censored at last known alive date prior to crossover.
Time Frame: From date of randomization until date of death from any cause, assessed up approximately 165 months
Population: Intent-to-Treat (ITT) population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 326 | 326
Months | 30.0 [24.2 to NA] — Not estimable due to insufficient number of participants with events | 38.3 [31.0 to NA] — Not estimable due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); Overall Survival (OS) (IIT population); Test type: Other; Hazard Ratio (HR) = 1.3786, 95% CI 2-sided [1.0246 to 1.8549] — Stratified HR for LTax/L versus TTax/T

4. Secondary Outcome: Overall Survival (OS) (Central HER2+ Population)
Description: as for outcome 3
Time Frame: From date of randomization until date of death from any cause, assessed up approximately 165 months
Population: Centrally-confirmed HER2 positive population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 270 | 267
Months | 30.0 [24.2 to NA] — Not estimable due to insufficient number of participants with events | NA [NA to NA] — Not estimable due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); Overall Survival (OS) (Central HER2+ population); Test type: Other; Hazard Ratio (HR) = 1.5818, 95% CI 2-sided [1.1181 to 2.2379] — Stratified HR for LTax/L versus TTax/T

5. Secondary Outcome: Incidence of Central Nervous System (CNS) Metastasis at First Progression (IIT Population)
Description: The incidence of Central Nervous System (CNS) metastasis at first progression was defined as the ratio of the number of subjects with CNS metastasis at progression over the total number of subjects.
Time Frame: From date of randomization to CNS metastases at time of first progression, assessed up approximately 45 months
Population: Participants in the Intent-to-Treat (ITT) population with available data for the outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Crossed Over to Trastuzumab (TTax/T) After IA Results: Crossed over to Trastuzumab (TTax/T) after IA results
- Overall TTax/T: Overall TTax/T
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T) | Crossed Over to Trastuzumab (TTax/T) After IA Results | Overall TTax/T
Number analyzed (Participants) | 326 | 326 | 5 | 331
Participants
  Subject had CNS metastasis at first progression = Yes: number analyzed (Participants) | 268 | 236 | 5 | 241
  Subject had CNS metastasis at first progression = Yes | 47 | 55 | 1 | 56
  Subject had CNS metastasis at first progression = No: number analyzed (Participants) | 268 | 236 | 5 | 241
  Subject had CNS metastasis at first progression = No | 155 | 119 | 4 | 123
  Subject had CNS metastasis at first progression = Unknown: number analyzed (Participants) | 268 | 236 | 5 | 241
  Subject had CNS metastasis at first progression = Unknown | 66 | 62 | 0 | 62

6. Secondary Outcome: Incidence of Central Nervous System (CNS) Metastasis at First Progression (Central HER2+ Population)
Description: as for outcome 5
Time Frame: From date of randomization to CNS metastases at time of first progression, assessed up approximately 45 months
Population: Participants in the centrally-confirmed HER2 positive population with available data for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T) | Crossed Over to Trastuzumab (TTax/T) After IA Results | Overall TTax/T
Number analyzed (Participants) | 270 | 267 | 4 | 271
Participants
  Subject had CNS metastasis at first progression = Yes: number analyzed (Participants) | 224 | 186 | 4 | 190
  Subject had CNS metastasis at first progression = Yes | 43 | 50 | 1 | 51
  Subject had CNS metastasis at first progression = No: number analyzed (Participants) | 224 | 186 | 4 | 190
  Subject had CNS metastasis at first progression = No | 128 | 92 | 3 | 95
  Subject had CNS metastasis at first progression = Unknown: number analyzed (Participants) | 224 | 186 | 4 | 190
  Subject had CNS metastasis at first progression = Unknown | 53 | 44 | 0 | 44

7. Secondary Outcome: Time to Central Nervous System (CNS) Metastasis (IIT Population)
Description: Time to Central Nervous System (CNS) metastasis was defined as the time from randomization until disease progression where CNS metastasis was documented at the time of first breast cancer progression. Subjects who crossed over the treatment to Trastuzumab (TTax/T) after interim analysis, were censored at RECIST assessment prior to crossover.
Time Frame: From date of randomization to CNS metastases at time of first progression, assessed up approximately 45 months
Population: Participants in the Intent-to-Treat (ITT) population with available data for the outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 47 | 55
Months | NA [NA to NA] — Not estimable due to number of events censored | NA [NA to NA] — Not estimable due to number of events censored
Statistical Analysis 1: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); Time to Central Nervous System (CNS) metastasis (IIT population); Test type: Other; Hazard Ratio (HR) = 1.0916, 95% CI 2-sided [0.7271 to 1.6389] — Stratified HR for LTax/L versus TTax/T

8. Secondary Outcome: Time to Central Nervous System (CNS) Metastasis (Central HER2+ Population)
Description: as for outcome 7
Time Frame: From date of randomization to CNS metastases at time of first progression, assessed up approximately 45 months
Population: Participants in the centrally-confirmed HER2 positive population with available data for the outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 43 | 50
Months | NA [25.4 to NA] — Not estimable due to number of events censored | NA [27.7 to NA] — Not estimable due to number of events censored
Statistical Analysis 1: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); Time to Central Nervous System (CNS) metastasis (Central HER2+ population); Test type: Other; Hazard Ratio (HR) = 1.0951, 95% CI 2-sided [0.7144 to 1.6787] — Stratified HR for LTax/L versus TTax/T

9. Secondary Outcome: Overall Response Rate (ORR) (IIT Population)
Description: Overall Response Rate (ORR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). The ORR was calculated from the Investigator's assessment of response based on RECIST 1.1. Subjects with an unknown or missing response were treated as non-responders; i.e., they were included in the denominator when calculating the percentages.
  Per Response Evaluation Criteria In Solid Tumors (RECIST v1.1) for target lesions and assessed by MRI:
  * Complete Response (CR): Disappearance of all target and non-target lesions.
  * Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as a reference the Baseline sum LD.
  * Overall Response (OR): CR + PR.
Time Frame: From date of randomization until date of progression or date of death from any cause, whichever comes first, assessed up approximately 45 months
Population: Intent-to-Treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 326 | 326
Percentage of Participants | 64.2 [58.0 to 70.1] | 63.3 [57.3 to 69.1]

10. Secondary Outcome: Overall Response Rate (ORR) (Central HER2+ Population)
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Centrally-confirmed HER2 positive population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 270 | 267
Percentage of Participants | 66.7 [60.0 to 72.9] | 67.4 [60.8 to 73.5]

11. Secondary Outcome: Clinical Benefit Response (CBR) (IIT Population)
Description: Clinical Benefit Response (CBR) was defined as the percentage with evidence of Complete Response (CR), Partial Response (PR) (participants with at least 1 measurable lesion at baseline), or maintaining Stable Disease (SD) for at least 24 weeks (all subjects, with or without measurable disease at baseline) while on study, according to the investigator assessment of response per RECIST 1.1 criteria. Participants were considered to be positive (Yes) for CBR if they experienced any CR or PR for any duration prior to progressive disease. Participants were considered to be negative (No) for CBR if they had progressive disease prior to Week 24 without prior confirmed CR or PR.
Time Frame: as for outcome 9
Population: Intent-to-Treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 326 | 326
Percentage of Participants | 60.4 [54.9 to 65.8] | 62.0 [56.5 to 67.3]

12. Secondary Outcome: Clinical Benefit Response (CBR) (Central HER2+ Population)
Description: as for outcome 11
Time Frame: as for outcome 9
Population: Centrally-confirmed HER2 positive population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 270 | 267
Percentage of Participants | 61.1 [55.0 to 67.0] | 65.2 [59.1 to 70.9]

13. Secondary Outcome: Time to Response (TTR) (IIT Population)
Description: Time to Response was defined as the time from randomization to the earliest date of Complete Response (CR) or Partial Response (PR). The event of first response was the first CR or PR; censoring was at PD date for those who progressed or at the last RECIST date if no progression occurred.
Time Frame: From date of randomization until date of first response, assessed up approximately 45 months
Population: Intent-to-Treat (ITT) Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 326 | 326
Months | 2.9 [2.8 to 3.0] | 2.9 [2.8 to 3.0]
Statistical Analysis 1: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); Time to Response (TTR) (IIT population); Test type: Other; Hazard Ratio (HR) = 1.0091, 95% CI 2-sided [0.8090 to 1.2586] — Stratified HR for LTax/L versus TTax/T

14. Secondary Outcome: Time to Response (TTR) (Central HER2+ Population)
Description: as for outcome 13
Time Frame: as for outcome 9
Population: Centrally-confirmed HER2 positive population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 270 | 267
Months | 2.9 [2.8 to 3.0] | 2.9 [2.8 to 3.0]
Statistical Analysis 1: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); Time to Response (TTR) (Central HER2+ population); Test type: Other; Hazard Ratio (HR) = 0.9573, 95% CI 2-sided [0.7544 to 1.2148] — Stratified HR for LTax/L versus TTax/T

15. Secondary Outcome: Duration of Response (DoR) (IIT Population)
Description: Duration of Response (DOR) was defined as the duration between the date of first documented Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) and the date of first documented sign of Progressive Disease or Death, with censoring at the last RECIST date if no progression occurred.
Time Frame: From first documented evidence of CR or PR (the response prior to confirmation) until time of documented disease progression or death due to any cause, whichever comes first, assessed up approximately 165 months
Population: Intent-to-Treat (ITT) Population. Subset of participants with at least one measurable lesion at baseline achieving either a confirmed complete response (CR) or partial response (PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 165 | 171
Months | 8.3 [7.6 to 9.4] | 11.1 [9.6 to 12.5]
Statistical Analysis 1: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); Duration of Response (DoR) (IIT population); Test type: Other; Hazard Ratio (HR) = 1.4866, 95% CI 2-sided [1.1479 to 1.9251] — Stratified HR for LTax/L versus TTax/T

16. Secondary Outcome: Duration of Response (DoR) (Central HER2+ Population)
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Centrally-confirmed HER2 positive population. Subset of participants with at least one measurable lesion at baseline achieving either a confirmed complete response (CR) or partial response (PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 144 | 151
Months | 8.3 [7.2 to 9.9] | 11.1 [10.6 to 13.8]
Statistical Analysis 1: Comparison: Lapatinib (LTax/L) vs Trastuzumab (TTax/T); Duration of Response (DoR) (Central HER2+ population); Test type: Other; Hazard Ratio (HR) = 1.5594, 95% CI 2-sided [1.1767 to 2.0666] — Stratified HR for LTax/L versus TTax/T

17. Secondary Outcome: EORTC QLQ-C30 Global Score at 12 Weeks
Description: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQC-30) is a questionnaire developed to assess the quality of life of cancer patients. The global score ranges from 0-100, with higher values representing a better quality of life.
Time Frame: Week 12
Population: Participants in the safety population with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: Score on global scale
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 260 | 266
Score on global scale | 61.67 (20.93) | 64.41 (20.18)

18. Secondary Outcome: Number of Participants Achieving European Quality of Life (EuroQol) - 5 Domain (EQ-5D) Score (Canadian and Australian Centers Only)
Description: The European Quality of Life (EuroQol) - 5 Domain (EQ-5D) self-administered questionnaire consists of two pages comprising the EQ-5D descriptive system and the EQ Visual Analogue Scale (VAS). The EQ-5D descriptive system comprises five dimensions of health (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and each dimension comprises three levels (no problems, some problems, extreme problems, unable to perform the activity).
Time Frame: Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 120, Week 144
Population: Safety Set - Canadian and Australian centers only. At each time point, only participants with a value at both Baseline and post-baseline time points were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 56 | 49
Participants
  Mobility @ Week 12: number analyzed (Participants) | 46 | 36
  Mobility @ Week 12: No Problems | 29 | 27
  Mobility @ Week 12: Some problems | 16 | 9
  Mobility @ Week 12: Unable to perform the activity | 1 | 0
  Mobility @ Week 12: Missing | 0 | 0
  Mobility @ Week 12: Not Done | 0 | 0
  Self-Care @ Week 12: number analyzed (Participants) | 46 | 36
  Self-Care @ Week 12: No Problems | 41 | 32
  Self-Care @ Week 12: Some problems | 4 | 2
  Self-Care @ Week 12: Unable to perform the activity | 1 | 1
  Self-Care @ Week 12: Missing | 0 | 1
  Self-Care @ Week 12: Not Done | 0 | 0
  Usual Activities @ Week 12: number analyzed (Participants) | 46 | 36
  Usual Activities @ Week 12: No Problems | 16 | 22
  Usual Activities @ Week 12: Some problems | 25 | 13
  Usual Activities @ Week 12: Unable to perform the activity | 5 | 1
  Usual Activities @ Week 12: Missing | 0 | 0
  Usual Activities @ Week 12: Not Done | 0 | 0
  Pain/Discomfort @ Week 12: number analyzed (Participants) | 46 | 36
  Pain/Discomfort @ Week 12: No Problems | 16 | 16
  Pain/Discomfort @ Week 12: Some problems | 28 | 20
  Pain/Discomfort @ Week 12: Unable to perform the activity | 1 | 0
  Pain/Discomfort @ Week 12: Missing | 1 | 0
  Pain/Discomfort @ Week 12: Not Done | 0 | 0
  Anxiety/Depression @ Week 12: number analyzed (Participants) | 46 | 36
  Anxiety/Depression @ Week 12: No Problems | 24 | 22
  Anxiety/Depression @ Week 12: Some problems | 20 | 14
  Anxiety/Depression @ Week 12: Unable to perform the activity | 2 | 0
  Anxiety/Depression @ Week 12: Missing | 0 | 0
  Anxiety/Depression @ Week 12: Not Done | 0 | 0
  Mobility @ Week 24: number analyzed (Participants) | 41 | 34
  Mobility @ Week 24: No Problems | 26 | 20
  Mobility @ Week 24: Some problems | 14 | 14
  Mobility @ Week 24: Unable to perform the activity | 1 | 0
  Mobility @ Week 24: Missing | 0 | 0
  Mobility @ Week 24: Not Done | 0 | 0
  Self-Care @ Week 24: number analyzed (Participants) | 41 | 34
  Self-Care @ Week 24: No Problems | 38 | 31
  Self-Care @ Week 24: Some problems | 3 | 3
  Self-Care @ Week 24: Unable to perform the activity | 0 | 0
  Self-Care @ Week 24: Missing | 0 | 0
  Self-Care @ Week 24: Not Done | 0 | 0
  Usual Activities @ Week 24: number analyzed (Participants) | 41 | 34
  Usual Activities @ Week 24: No Problems | 18 | 18
  Usual Activities @ Week 24: Some problems | 22 | 14
  Usual Activities @ Week 24: Unable to perform the activity | 1 | 2
  Usual Activities @ Week 24: Missing | 0 | 0
  Usual Activities @ Week 24: Not Done | 0 | 0
  Pain/Discomfort @ Week 24: number analyzed (Participants) | 41 | 34
  Pain/Discomfort @ Week 24: No Problems | 10 | 12
  Pain/Discomfort @ Week 24: Some problems | 30 | 21
  Pain/Discomfort @ Week 24: Unable to perform the activity | 1 | 1
  Pain/Discomfort @ Week 24: Missing | 0 | 0
  Pain/Discomfort @ Week 24: Not Done | 0 | 0
  Anxiety/Depression @ Week 24: number analyzed (Participants) | 41 | 34
  Anxiety/Depression @ Week 24: No Problems | 23 | 18
  Anxiety/Depression @ Week 24: Some problems | 18 | 15
  Anxiety/Depression @ Week 24: Unable to perform the activity | 0 | 1
  Anxiety/Depression @ Week 24: Missing | 0 | 0
  Anxiety/Depression @ Week 24: Not Done | 0 | 0
  Mobility @ Week 36: number analyzed (Participants) | 31 | 31
  Mobility @ Week 36: No Problems | 21 | 26
  Mobility @ Week 36: Some problems | 10 | 5
  Mobility @ Week 36: Unable to perform the activity | 0 | 0
  Mobility @ Week 36: Missing | 0 | 0
  Mobility @ Week 36: Not Done | 0 | 0
  Self-Care @ Week 36: number analyzed (Participants) | 31 | 31
  Self-Care @ Week 36: No Problems | 28 | 30
  Self-Care @ Week 36: Some problems | 2 | 1
  Self-Care @ Week 36: Unable to perform the activity | 0 | 0
  Self-Care @ Week 36: Missing | 0 | 0
  Self-Care @ Week 36: Not Done | 1 | 0
  Usual Activities @ Week 36: number analyzed (Participants) | 31 | 31
  Usual Activities @ Week 36: No Problems | 17 | 16
  Usual Activities @ Week 36: Some problems | 13 | 14
  Usual Activities @ Week 36: Unable to perform the activity | 0 | 1
  Usual Activities @ Week 36: Missing | 0 | 0
  Usual Activities @ Week 36: Not Done | 1 | 0
  Pain/Discomfort @ Week 36: number analyzed (Participants) | 31 | 31
  Pain/Discomfort @ Week 36: No Problems | 9 | 13
  Pain/Discomfort @ Week 36: Some problems | 18 | 16
  Pain/Discomfort @ Week 36: Unable to perform the activity | 3 | 1
  Pain/Discomfort @ Week 36: Missing | 0 | 1
  Pain/Discomfort @ Week 36: Not Done | 1 | 0
  Anxiety/Depression @ Week 36: number analyzed (Participants) | 31 | 31
  Anxiety/Depression @ Week 36: No Problems | 18 | 18
  Anxiety/Depression @ Week 36: Some problems | 12 | 13
  Anxiety/Depression @ Week 36: Unable to perform the activity | 0 | 0
  Anxiety/Depression @ Week 36: Missing | 0 | 0
  Anxiety/Depression @ Week 36: Not Done | 1 | 0
  Mobility @ Week 48: number analyzed (Participants) | 18 | 27
  Mobility @ Week 48: No Problems | 14 | 18
  Mobility @ Week 48: Some problems | 4 | 9
  Mobility @ Week 48: Unable to perform the activity | 0 | 0
  Mobility @ Week 48: Missing | 0 | 0
  Mobility @ Week 48: Not Done | 0 | 0
  Self-Care @ Week 48: number analyzed (Participants) | 18 | 27
  Self-Care @ Week 48: No Problems | 18 | 26
  Self-Care @ Week 48: Some problems | 0 | 1
  Self-Care @ Week 48: Unable to perform the activity | 0 | 0
  Self-Care @ Week 48: Missing | 0 | 0
  Self-Care @ Week 48: Not Done | 0 | 0
  Usual Activities @ Week 48: number analyzed (Participants) | 18 | 27
  Usual Activities @ Week 48: No Problems | 15 | 16
  Usual Activities @ Week 48: Some problems | 3 | 11
  Usual Activities @ Week 48: Unable to perform the activity | 0 | 0
  Usual Activities @ Week 48: Missing | 0 | 0
  Usual Activities @ Week 48: Not Done | 0 | 0
  Pain/Discomfort @ Week 48: number analyzed (Participants) | 18 | 27
  Pain/Discomfort @ Week 48: No Problems | 6 | 12
  Pain/Discomfort @ Week 48: Some problems | 11 | 14
  Pain/Discomfort @ Week 48: Unable to perform the activity | 1 | 0
  Pain/Discomfort @ Week 48: Missing | 0 | 1
  Pain/Discomfort @ Week 48: Not Done | 0 | 0
  Anxiety/Depression @ Week 48: number analyzed (Participants) | 18 | 27
  Anxiety/Depression @ Week 48: No Problems | 10 | 20
  Anxiety/Depression @ Week 48: Some problems | 7 | 6
  Anxiety/Depression @ Week 48: Unable to perform the activity | 0 | 1
  Anxiety/Depression @ Week 48: Missing | 1 | 0
  Anxiety/Depression @ Week 48: Not Done | 0 | 0
  Mobility @ Week 60: number analyzed (Participants) | 8 | 21
  Mobility @ Week 60: No Problems | 8 | 16
  Mobility @ Week 60: Some problems | 0 | 5
  Mobility @ Week 60: Unable to perform the activity | 0 | 0
  Mobility @ Week 60: Missing | 0 | 0
  Mobility @ Week 60: Not Done | 0 | 0
  Self-Care @ Week 60: number analyzed (Participants) | 8 | 21
  Self-Care @ Week 60: No Problems | 8 | 20
  Self-Care @ Week 60: Some problems | 0 | 1
  Self-Care @ Week 60: Unable to perform the activity | 0 | 0
  Self-Care @ Week 60: Missing | 0 | 0
  Self-Care @ Week 60: Not Done | 0 | 0
  Usual Activities @ Week 60: number analyzed (Participants) | 8 | 21
  Usual Activities @ Week 60: No Problems | 7 | 12
  Usual Activities @ Week 60: Some problems | 1 | 7
  Usual Activities @ Week 60: Unable to perform the activity | 0 | 2
  Usual Activities @ Week 60: Missing | 0 | 0
  Usual Activities @ Week 60: Not Done | 0 | 0
  Pain/Discomfort @ Week 60: number analyzed (Participants) | 8 | 21
  Pain/Discomfort @ Week 60: No Problems | 5 | 11
  Pain/Discomfort @ Week 60: Some problems | 3 | 8
  Pain/Discomfort @ Week 60: Unable to perform the activity | 0 | 2
  Pain/Discomfort @ Week 60: Missing | 0 | 0
  Pain/Discomfort @ Week 60: Not Done | 0 | 0
  Anxiety/Depression @ Week 60: number analyzed (Participants) | 8 | 21
  Anxiety/Depression @ Week 60: No Problems | 5 | 12
  Anxiety/Depression @ Week 60: Some problems | 3 | 9
  Anxiety/Depression @ Week 60: Unable to perform the activity | 0 | 0
  Anxiety/Depression @ Week 60: Missing | 0 | 0
  Anxiety/Depression @ Week 60: Not Done | 0 | 0
  Mobility @ Week 72: number analyzed (Participants) | 8 | 15
  Mobility @ Week 72: No Problems | 7 | 13
  Mobility @ Week 72: Some problems | 1 | 2
  Mobility @ Week 72: Unable to perform the activity | 0 | 0
  Mobility @ Week 72: Missing | 0 | 0
  Mobility @ Week 72: Not Done | 0 | 0
  Self-Care @ Week 72: number analyzed (Participants) | 8 | 15
  Self-Care @ Week 72: No Problems | 8 | 15
  Self-Care @ Week 72: Some problems | 0 | 0
  Self-Care @ Week 72: Unable to perform the activity | 0 | 0
  Self-Care @ Week 72: Missing | 0 | 0
  Self-Care @ Week 72: Not Done | 0 | 0
  Usual Activities @ Week 72: number analyzed (Participants) | 8 | 15
  Usual Activities @ Week 72: No Problems | 7 | 8
  Usual Activities @ Week 72: Some problems | 1 | 7
  Usual Activities @ Week 72: Unable to perform the activity | 0 | 0
  Usual Activities @ Week 72: Missing | 0 | 0
  Usual Activities @ Week 72: Not Done | 0 | 0
  Pain/Discomfort @ Week 72: number analyzed (Participants) | 8 | 15
  Pain/Discomfort @ Week 72: No Problems | 6 | 9
  Pain/Discomfort @ Week 72: Some problems | 2 | 6
  Pain/Discomfort @ Week 72: Unable to perform the activity | 0 | 0
  Pain/Discomfort @ Week 72: Missing | 0 | 0
  Pain/Discomfort @ Week 72: Not Done | 0 | 0
  Anxiety/Depression @ Week 72: number analyzed (Participants) | 8 | 15
  Anxiety/Depression @ Week 72: No Problems | 4 | 8
  Anxiety/Depression @ Week 72: Some problems | 4 | 6
  Anxiety/Depression @ Week 72: Unable to perform the activity | 0 | 1
  Anxiety/Depression @ Week 72: Missing | 0 | 0
  Anxiety/Depression @ Week 72: Not Done | 0 | 0
  Mobility @ Week 84: number analyzed (Participants) | 6 | 8
  Mobility @ Week 84: No Problems | 5 | 6
  Mobility @ Week 84: Some problems | 1 | 2
  Mobility @ Week 84: Unable to perform the activity | 0 | 0
  Mobility @ Week 84: Missing | 0 | 0
  Mobility @ Week 84: Not Done | 0 | 0
  Self-Care @ Week 84: number analyzed (Participants) | 6 | 8
  Self-Care @ Week 84: No Problems | 6 | 8
  Self-Care @ Week 84: Some problems | 0 | 0
  Self-Care @ Week 84: Unable to perform the activity | 0 | 0
  Self-Care @ Week 84: Missing | 0 | 0
  Self-Care @ Week 84: Not Done | 0 | 0
  Usual Activities @ Week 84: number analyzed (Participants) | 6 | 8
  Usual Activities @ Week 84: No Problems | 5 | 5
  Usual Activities @ Week 84: Some problems | 1 | 2
  Usual Activities @ Week 84: Unable to perform the activity | 0 | 1
  Usual Activities @ Week 84: Missing | 0 | 0
  Usual Activities @ Week 84: Not Done | 0 | 0
  Pain/Discomfort @ Week 84: number analyzed (Participants) | 6 | 8
  Pain/Discomfort @ Week 84: No Problems | 4 | 2
  Pain/Discomfort @ Week 84: Some problems | 2 | 6
  Pain/Discomfort @ Week 84: Unable to perform the activity | 0 | 0
  Pain/Discomfort @ Week 84: Missing | 0 | 0
  Pain/Discomfort @ Week 84: Not Done | 0 | 0
  Anxiety/Depression @ Week 84: number analyzed (Participants) | 6 | 8
  Anxiety/Depression @ Week 84: No Problems | 3 | 4
  Anxiety/Depression @ Week 84: Some problems | 3 | 4
  Anxiety/Depression @ Week 84: Unable to perform the activity | 0 | 0
  Anxiety/Depression @ Week 84: Missing | 0 | 0
  Anxiety/Depression @ Week 84: Not Done | 0 | 0
  Mobility @ Week 96: number analyzed (Participants) | 5 | 5
  Mobility @ Week 96: No Problems | 5 | 3
  Mobility @ Week 96: Some problems | 0 | 2
  Mobility @ Week 96: Unable to perform the activity | 0 | 0
  Mobility @ Week 96: Missing | 0 | 0
  Mobility @ Week 96: Not Done | 0 | 0
  Self-Care @ Week 96: number analyzed (Participants) | 5 | 5
  Self-Care @ Week 96: No Problems | 5 | 5
  Self-Care @ Week 96: Some problems | 0 | 0
  Self-Care @ Week 96: Unable to perform the activity | 0 | 0
  Self-Care @ Week 96: Missing | 0 | 0
  Self-Care @ Week 96: Not Done | 0 | 0
  Usual Activities @ Week 96: number analyzed (Participants) | 5 | 5
  Usual Activities @ Week 96: No Problems | 3 | 3
  Usual Activities @ Week 96: Some problems | 2 | 2
  Usual Activities @ Week 96: Unable to perform the activity | 0 | 0
  Usual Activities @ Week 96: Missing | 0 | 0
  Usual Activities @ Week 96: Not Done | 0 | 0
  Pain/Discomfort @ Week 96: number analyzed (Participants) | 5 | 5
  Pain/Discomfort @ Week 96: No Problems | 2 | 1
  Pain/Discomfort @ Week 96: Some problems | 2 | 4
  Pain/Discomfort @ Week 96: Unable to perform the activity | 1 | 0
  Pain/Discomfort @ Week 96: Missing | 0 | 0
  Pain/Discomfort @ Week 96: Not Done | 0 | 0
  Anxiety/Depression @ Week 96: number analyzed (Participants) | 5 | 5
  Anxiety/Depression @ Week 96: No Problems | 1 | 3
  Anxiety/Depression @ Week 96: Some problems | 4 | 2
  Anxiety/Depression @ Week 96: Unable to perform the activity | 0 | 0
  Anxiety/Depression @ Week 96: Missing | 0 | 0
  Anxiety/Depression @ Week 96: Not Done | 0 | 0
  Mobility @ Week 120: number analyzed (Participants) | 4 | 3
  Mobility @ Week 120: No Problems | 4 | 2
  Mobility @ Week 120: Some problems | 0 | 1
  Mobility @ Week 120: Unable to perform the activity | 0 | 0
  Mobility @ Week 120: Missing | 0 | 0
  Mobility @ Week 120: Not Done | 0 | 0
  Self-Care @ Week 120: number analyzed (Participants) | 4 | 3
  Self-Care @ Week 120: No Problems | 4 | 3
  Self-Care @ Week 120: Some problems | 0 | 0
  Self-Care @ Week 120: Unable to perform the activity | 0 | 0
  Self-Care @ Week 120: Missing | 0 | 0
  Self-Care @ Week 120: Not Done | 0 | 0
  Usual Activities @ Week 120: number analyzed (Participants) | 4 | 3
  Usual Activities @ Week 120: No Problems | 4 | 2
  Usual Activities @ Week 120: Some problems | 0 | 1
  Usual Activities @ Week 120: Unable to perform the activity | 0 | 0
  Usual Activities @ Week 120: Missing | 0 | 0
  Usual Activities @ Week 120: Not Done | 0 | 0
  Pain/Discomfort @ Week 120: number analyzed (Participants) | 4 | 3
  Pain/Discomfort @ Week 120: No Problems | 3 | 2
  Pain/Discomfort @ Week 120: Some problems | 1 | 1
  Pain/Discomfort @ Week 120: Unable to perform the activity | 0 | 0
  Pain/Discomfort @ Week 120: Missing | 0 | 0
  Pain/Discomfort @ Week 120: Not Done | 0 | 0
  Anxiety/Depression @ Week 120: number analyzed (Participants) | 4 | 3
  Anxiety/Depression @ Week 120: No Problems | 1 | 3
  Anxiety/Depression @ Week 120: Some problems | 3 | 0
  Anxiety/Depression @ Week 120: Unable to perform the activity | 0 | 0
  Anxiety/Depression @ Week 120: Missing | 0 | 0
  Anxiety/Depression @ Week 120: Not Done | 0 | 0
  Mobility @ Week 144: number analyzed (Participants) | 1 | 1
  Mobility @ Week 144: No Problems | 1 | 1
  Mobility @ Week 144: Some problems | 0 | 0
  Mobility @ Week 144: Unable to perform the activity | 0 | 0
  Mobility @ Week 144: Missing | 0 | 0
  Mobility @ Week 144: Not Done | 0 | 0
  Self-Care @ Week 144: number analyzed (Participants) | 1 | 1
  Self-Care @ Week 144: No Problems | 1 | 1
  Self-Care @ Week 144: Some problems | 0 | 0
  Self-Care @ Week 144: Unable to perform the activity | 0 | 0
  Self-Care @ Week 144: Missing | 0 | 0
  Self-Care @ Week 144: Not Done | 0 | 0
  Usual Activities @ Week 144: number analyzed (Participants) | 1 | 1
  Usual Activities @ Week 144: No Problems | 1 | 1
  Usual Activities @ Week 144: Some problems | 0 | 0
  Usual Activities @ Week 144: Unable to perform the activity | 0 | 0
  Usual Activities @ Week 144: Missing | 0 | 0
  Usual Activities @ Week 144: Not Done | 0 | 0
  Pain/Discomfort @ Week 144: number analyzed (Participants) | 1 | 1
  Pain/Discomfort @ Week 144: No Problems | 1 | 1
  Pain/Discomfort @ Week 144: Some problems | 0 | 0
  Pain/Discomfort @ Week 144: Unable to perform the activity | 0 | 0
  Pain/Discomfort @ Week 144: Missing | 0 | 0
  Pain/Discomfort @ Week 144: Not Done | 0 | 0
  Anxiety/Depression @ Week 144: number analyzed (Participants) | 1 | 1
  Anxiety/Depression @ Week 144: No Problems | 0 | 1
  Anxiety/Depression @ Week 144: Some problems | 1 | 0
  Anxiety/Depression @ Week 144: Unable to perform the activity | 0 | 0
  Anxiety/Depression @ Week 144: Missing | 0 | 0
  Anxiety/Depression @ Week 144: Not Done | 0 | 0

19. Secondary Outcome: Change From Baseline in the EQ-VAS Score (Canadian and Australian Centers Only)
Description: The European Quality of Life (EuroQol) - 5 Domain (EQ-5D) self-administered questionnaire consists of two pages comprising the EQ-5D descriptive system and the EQ Visual Analogue Scale (VAS). The EQ VAS records the patient's self-rated health on a vertical visual analogue 0-100 scale, where the endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0).
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 120, Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 55 | 43
Score on a scale
  Week 12: number analyzed (Participants) | 46 | 36
  Week 12 | 1.6 (17.16) | 7.0 (19.30)
  Week 24: number analyzed (Participants) | 41 | 34
  Week 24 | -1.5 (21.98) | 1.3 (21.56)
  Week 36: number analyzed (Participants) | 31 | 31
  Week 36 | 0.4 (21.86) | 5.9 (22.53)
  Week 48: number analyzed (Participants) | 18 | 27
  Week 48 | 5.2 (23.17) | 6.5 (25.37)
  Week 60: number analyzed (Participants) | 8 | 21
  Week 60 | 5.8 (10.51) | 7.9 (28.29)
  Week 72: number analyzed (Participants) | 8 | 15
  Week 72 | 10.1 (7.36) | 11.8 (29.96)
  Week 84: number analyzed (Participants) | 6 | 8
  Week 84 | 5.2 (6.46) | 4.9 (25.08)
  Week 96: number analyzed (Participants) | 5 | 5
  Week 96 | 3.0 (19.90) | -10.0 (10.80)
  Week 120: number analyzed (Participants) | 4 | 3
  Week 120 | 10.3 (5.91) | -11.0 (13.11)
  Week 144: number analyzed (Participants) | 1 | 1
  Week 144 | 13.0 (NA) — Only 1 participant analyzed | 4.0 (NA) — Only 1 participant analyzed

20. Secondary Outcome: Number of Participants With Healthcare Utilization (Canadian and Australian Centers Only)
Description: The measures of healthcare resource utilization collected were categorized: hospitalization/inpatient visit, Institutionalized, Outpatient visit.
Time Frame: From date of randomization till 28 days safety follow-up, assessed up to 40 months
Population: Safety Set - Canadian and Australian centers only
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 56 | 49
Participants
  Hospitalization/Inpatient visit | 29 | 17
  Institutionalized | 0 | 2
  Outpatient Visit | 52 | 45

21. Secondary Outcome: Number of Participant Hospitalized (Canadian and Australian Centers Only)
Description: The number of hospitalizations were categorized: >0 and =<2, >2 and =<4 and >4.
Time Frame: From date of randomization till 28 days safety follow-up, assessed up to 40 months
Population: Safety Set - Canadian and Australian centers only and for participants with Hospitalization/Inpatient visit
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 29 | 17
Participants
  > 0 and =< 2 | 27 | 16
  > 2 and =< 4 | 1 | 0
  > 4 | 1 | 1

22. Secondary Outcome: Total and Average Duration of Hospitalization (Canadian and Australian Centers Only)
Description: The total duration of hospitalization in days and average duration of each hospitalization in days were summarized using descriptive statistics.
Time Frame: From date of randomization till 28 days safety follow-up, assessed up to 40 months
Population: Safety Set - Canadian and Australian centers only and for participants with Hospitalization/Inpatient visit
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 29 | 17
Days
  Total duration of hospitalization | 10.38 (10.63) | 16.18 (38.63)
  Average duration of each hospitalization | 6.6 (5.46) | 6.5 (4.81)

23. Secondary Outcome: Reasons for Hospitalization (Canadian and Australian Centers Only)
Description: The reasons for hospitalization were categorized: Breast Cancer, Febrile Neutropenia, Infection, Other and Pneumonia.
Time Frame: From date of randomization till 28 days safety follow-up, assessed up to 40 months
Population: Safety Set - Canadian and Australian centers only and for participants with Hospitalization/Inpatient visit
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 29 | 17
Participants
  Breast Cancer | 3 | 3
  Febrile neutropenia | 10 | 1
  Infection | 5 | 4
  Other | 14 | 9
  Pneumonia | 2 | 1

24. Secondary Outcome: Type of Ward (Hospital Unit) (Canadian and Australian Centers Only)
Description: The type of ward (hospital unit) were categorized: general ward, intensive care unit, oncology ward, rehabilitation unit and other.
Time Frame: From date of randomization till 28 days safety follow-up, assessed up to 40 months
Population: Safety Set - Canadian and Australian centers only and for participants with Hospitalization/Inpatient visit
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 29 | 17
Participants
  General ward | 12 | 9
  Intensive care unit | 1 | 1
  Oncology ward | 13 | 9
  Other | 6 | 3
  Rehabilitation unit | 0 | 1

25. Secondary Outcome: Discharge Destinations (Canadian and Australian Centers Only)
Description: The discharge destinations were categorized: died, home, rehabilitation facility and transfer to other hospital.
Time Frame: From date of randomization till 28 days safety follow-up, assessed up to 40 months
Population: Safety Set - Canadian and Australian centers only and for participants with Hospitalization/Inpatient visit
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 29 | 17
Participants
  Died | 1 | 1
  Home | 26 | 14
  Rehabilitation facility | 0 | 1
  Transfer to other hospital | 1 | 1
  Unknwon/missing | 1 | 0

26. Secondary Outcome: Estrogen Receptor (ER) and Progesterone Receptor (PgR) Status
Description: Immunohistochemistry (IHC) analysis of estrogen receptor (ER) and progesterone receptor (PgR) were performed as part of the mandatory central laboratory testing for protocol-specified biomarkers.
Time Frame: Up to approximately 39 months
Population: Intent-to-Treat (ITT) population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Lapatinib (LTax/L) | Trastuzumab (TTax/T)
Number analyzed (Participants) | 326 | 326
Percentage of Participants
  estrogen receptor (ER) positive | 65 | 64
  progesterone receptor (PgR) negative | 58 | 63

27. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from day of participant's informed consent to the day before first dose of study medication.
  On-treatment deaths were collected from first dose of study medication to 28 days after last dose of study medication (on-treatment), up to approximately 165 months.
  Deaths were collected in the post treatment survival follow up from 29 days after last dose of study medication until the end of the study, up to approximately 166 months.
Time Frame: Pre-treatment deaths: Up to 1 month prior to treatment. On-treatment deaths: Up to 165 months. Post-treatment deaths: up to 166 months.
Population: Intent-to-Treat (ITT) Population.
Measure: Count of Participants; unit: Participants
Groups:
- Lapatinib (LTax/L) - All Participants: Lapatinib 1250 mg once daily. Taxane based chemotherapy: Paclitaxel 80 mg/m2 IV once weekly (Days 1, 8, and 15 of a 4-week cycle) OR Docetaxel 75 mg/m2 IV once every 3 weeks (Day 1 of a 3-week cycle) plus G-CSF: according to institutional standards. Followed by Lapatinib 1500 mg once daily until disease progression.
- Lapatinib (LTax/L) - Crossed Over to Trastuzumab (TTax/T) After IA Results: Lapatinib (LTax/L) - Crossed over to Trastuzumab (TTax/T) after IA results: Participants initially randomized to Lapatinib (LTax/L) who crossed over to Trastuzumab (TTax/T) after Interim Analysis (IA) results
Arm/Group | Lapatinib (LTax/L) - All Participants | Trastuzumab (TTax/T) | Lapatinib (LTax/L) - Crossed Over to Trastuzumab (TTax/T) After IA Results
Number analyzed (Participants) | 326 | 326 | 5
Participants
  Pre-treatment deaths: number analyzed (Participants) | 326 | 326 | 0
  Pre-treatment deaths | 0 | 0 | 0
  On-treatment deaths: number analyzed (Participants) | 322 | 325 | 5
  On-treatment deaths | 21 | 13 | 0
  Post-treatment deaths: number analyzed (Participants) | 301 | 312 | 5
  Post-treatment deaths | 82 | 73 | 0
  All deaths | 103 | 86 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of study medication until the last dose plus 28 days post-treat follow-up, assessed up to approximately 165 months. Deaths were recorded from study start date until end of survival follow-up phase (end of study), assessed up to approximately 166 months.
Description: Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival included patients who entered this period. All-cause Mortality was assessed for all participants enrolled in the study, while Serious and Other Adverse Events were assessed for all participants who received at least one dose of the study medication.
Groups:
- Lapatinib (LTax/L) - All Participants: Lapatinib (LTax/L) - All participants: Events up to 28 days post-treatment
- Trastuzumab (TTax/T): Trastuzumab (TTax/T): Events up to 28 days post-treatment
- Lapatinib (LTax/L) - Crossed Over to Trastuzumab (TTax/T) After IA Results: Lapatinib (LTax/L) - Crossed over to Trastuzumab (TTax/T) after IA results: Events up to 28 days post-treatment
- Lapatinib (LTax/L) - All Participants (Post-treatment): Lapatinib (LTax/L) - All participants (Post-treatment): Deaths in the post-treatment survival follow-up were not considered adverse events.
- Trastuzumab (TTax/T) (Post-treatment): Trastuzumab (TTax/T) (Post-treatment): Deaths in the post-treatment survival follow-up were not considered adverse events.
- Lapatinib (LTax/L) - Crossed Over to Trastuzumab (TTax/T) After IA Results (Post-treatment): Lapatinib (LTax/L) - Crossed over to Trastuzumab (TTax/T) after IA results: Deaths in the post-treatment survival follow-up were not considered adverse events.
Arm/Group | Lapatinib (LTax/L) - All Participants | Trastuzumab (TTax/T) | Lapatinib (LTax/L) - Crossed Over to Trastuzumab (TTax/T) After IA Results | Lapatinib (LTax/L) - All Participants (Post-treatment) | Trastuzumab (TTax/T) (Post-treatment) | Lapatinib (LTax/L) - Crossed Over to Trastuzumab (TTax/T) After IA Results (Post-treatment)
All-Cause Mortality (participants affected / at risk) | 21/326 | 13/326 | 0/5 | 82/301 | 73/312 | 0/5
Serious Adverse Events (participants affected / at risk) | 106/322 | 66/325 | 2/5 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 316/322 | 319/325 | 1/5 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib (LTax/L) - All Participants (N=322) | Trastuzumab (TTax/T) (N=325) | Lapatinib (LTax/L) - Crossed Over to Trastuzumab (TTax/T) After IA Results (N=5) | Lapatinib (LTax/L) - All Participants (Post-treatment) (N=0) | Trastuzumab (TTax/T) (Post-treatment) (N=0) | Lapatinib (LTax/L) - Crossed Over to Trastuzumab (TTax/T) After IA Results (Post-treatment) (N=0)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 3 | 0 | NA | NA | NA
Platelet disorder (Blood and lymphatic system disorders) | 0 | 1 | 0 | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0 | NA | NA | NA
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Chest pain (Cardiac disorders) | 1 | 1 | 0 | NA | NA | NA
Left ventricular dysfunction (Cardiac disorders) | 1 | 2 | 0 | NA | NA | NA
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Right ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 0 | NA | NA | NA
Sudden death (Cardiac disorders) | 1 | 1 | 0 | NA | NA | NA
Hypercalcaemia (Endocrine disorders) | 2 | 0 | 0 | NA | NA | NA
Hyperglycaemia (Endocrine disorders) | 2 | 2 | 0 | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | NA | NA | NA
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 23 | 5 | 0 | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Fistula of small intestine (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0 | NA | NA | NA
Gastrointestinal disorder (Gastrointestinal disorders) | 3 | 0 | 0 | NA | NA | NA
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Ileus (Gastrointestinal disorders) | 2 | 0 | 0 | NA | NA | NA
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Large intestine infection (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 6 | 4 | 0 | NA | NA | NA
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | NA | NA | NA
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | NA | NA | NA
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 12 | 3 | 0 | NA | NA | NA
Death (General disorders) | 2 | 2 | 0 | NA | NA | NA
Device related infection (General disorders) | 2 | 3 | 0 | NA | NA | NA
Fatigue (General disorders) | 5 | 1 | 0 | NA | NA | NA
Febrile neutropenia (General disorders) | 16 | 8 | 0 | NA | NA | NA
Pyrexia (General disorders) | 7 | 9 | 0 | NA | NA | NA
Ulcer (General disorders) | 1 | 0 | 0 | NA | NA | NA
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatobiliary disease (Hepatobiliary disorders) | 1 | 1 | 0 | NA | NA | NA
Hypersensitivity (Immune system disorders) | 2 | 3 | 0 | NA | NA | NA
Cystitis (Infections and infestations) | 5 | 1 | 0 | NA | NA | NA
Infection (Infections and infestations) | 10 | 2 | 0 | NA | NA | NA
Paronychia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Pneumonia (Infections and infestations) | 7 | 3 | 0 | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 4 | 0 | NA | NA | NA
Sinusitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Upper aerodigestive tract infection (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 4 | 1 | 0 | NA | NA | NA
Wound infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Fracture (Injury, poisoning and procedural complications) | 3 | 2 | 0 | NA | NA | NA
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Injection site reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Large intestine perforation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Alanine aminotransferase (Investigations) | 14 | 1 | 0 | NA | NA | NA
Aspartate aminotransferase (Investigations) | 7 | 1 | 0 | NA | NA | NA
Blood bilirubin (Investigations) | 7 | 0 | 0 | NA | NA | NA
Blood creatinine (Investigations) | 0 | 1 | 0 | NA | NA | NA
Haemoglobin (Investigations) | 1 | 2 | 0 | NA | NA | NA
Lipase (Investigations) | 0 | 1 | 0 | NA | NA | NA
Neutrophil count (Investigations) | 6 | 3 | 0 | NA | NA | NA
Weight decreased (Investigations) | 2 | 0 | 0 | NA | NA | NA
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 0 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | NA | NA | NA
Chills (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | NA | NA | NA
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Soft tissue infection (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Confusional state (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Multifocal motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Muscular weakness (Nervous system disorders) | 1 | 1 | 0 | NA | NA | NA
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | NA | NA | NA
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | NA | NA | NA
Kidney infection (Renal and urinary disorders) | 0 | 1 | 0 | NA | NA | NA
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Renal failure (Renal and urinary disorders) | 2 | 1 | 0 | NA | NA | NA
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 1 | 0 | NA | NA | NA
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | NA | NA | NA
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | NA | NA | NA
Skin infection (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | NA | NA | NA
Cerebral ischaemia (Vascular disorders) | 2 | 1 | 1 | NA | NA | NA
Disseminated intravascular coagulation (Vascular disorders) | 0 | 1 | 0 | NA | NA | NA
Embolism (Vascular disorders) | 5 | 4 | 0 | NA | NA | NA
Gastric haemorrhage (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Haematoma (Vascular disorders) | 0 | 1 | 0 | NA | NA | NA
Hypertension (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Syncope (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Uterine haemorrhage (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib (LTax/L) - All Participants (N=322) | Trastuzumab (TTax/T) (N=325) | Lapatinib (LTax/L) - Crossed Over to Trastuzumab (TTax/T) After IA Results (N=5) | Lapatinib (LTax/L) - All Participants (Post-treatment) (N=0) | Trastuzumab (TTax/T) (Post-treatment) (N=0) | Lapatinib (LTax/L) - Crossed Over to Trastuzumab (TTax/T) After IA Results (Post-treatment) (N=0)
Chest pain (Cardiac disorders) | 9 | 21 | 0 | NA | NA | NA
Left ventricular dysfunction (Cardiac disorders) | 9 | 25 | 0 | NA | NA | NA
Oedema peripheral (Cardiac disorders) | 86 | 113 | 0 | NA | NA | NA
Lacrimation increased (Eye disorders) | 26 | 37 | 0 | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 18 | 8 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 51 | 40 | 0 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 21 | 14 | 0 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 74 | 85 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 250 | 130 | 0 | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 19 | 12 | 0 | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 67 | 61 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 157 | 139 | 0 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 138 | 106 | 0 | NA | NA | NA
Taste disorder (Gastrointestinal disorders) | 55 | 51 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 92 | 75 | 0 | NA | NA | NA
Fatigue (General disorders) | 225 | 212 | 0 | NA | NA | NA
Pyrexia (General disorders) | 51 | 54 | 0 | NA | NA | NA
Hypersensitivity (Immune system disorders) | 30 | 45 | 1 | NA | NA | NA
Cystitis (Infections and infestations) | 15 | 22 | 0 | NA | NA | NA
Paronychia (Infections and infestations) | 29 | 11 | 0 | NA | NA | NA
Rhinitis (Infections and infestations) | 27 | 31 | 0 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 38 | 43 | 0 | NA | NA | NA
Gamma-glutamyltransferase (Investigations) | 20 | 10 | 0 | NA | NA | NA
Weight decreased (Investigations) | 29 | 14 | 0 | NA | NA | NA
Weight increased (Investigations) | 6 | 17 | 0 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 107 | 74 | 0 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 75 | 99 | 0 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 55 | 72 | 0 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 69 | 79 | 0 | NA | NA | NA
Chills (Musculoskeletal and connective tissue disorders) | 7 | 22 | 0 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 79 | 78 | 1 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 | 52 | 0 | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 22 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | 36 | 51 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 66 | 72 | 0 | NA | NA | NA
Multifocal motor neuropathy (Nervous system disorders) | 16 | 21 | 0 | NA | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Nervous system disorders) | 30 | 10 | 0 | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 168 | 165 | 0 | NA | NA | NA
Vision blurred (Nervous system disorders) | 16 | 17 | 0 | NA | NA | NA
Anxiety (Psychiatric disorders) | 34 | 34 | 0 | NA | NA | NA
Depressed mood (Psychiatric disorders) | 27 | 30 | 0 | NA | NA | NA
Dysphonia (Psychiatric disorders) | 8 | 21 | 0 | NA | NA | NA
Insomnia (Psychiatric disorders) | 65 | 72 | 0 | NA | NA | NA
Breast pain (Reproductive system and breast disorders) | 24 | 29 | 0 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 69 | 94 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 75 | 85 | 0 | NA | NA | NA
Influenza (Respiratory, thoracic and mediastinal disorders) | 23 | 30 | 0 | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 30 | 0 | NA | NA | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 30 | 21 | 0 | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 212 | 238 | 0 | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 59 | 40 | 0 | NA | NA | NA
Nail disorder (Skin and subcutaneous tissue disorders) | 129 | 88 | 0 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 38 | 0 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 192 | 127 | 0 | NA | NA | NA
Skin disorder (Skin and subcutaneous tissue disorders) | 25 | 20 | 0 | NA | NA | NA
Skin infection (Skin and subcutaneous tissue disorders) | 12 | 19 | 0 | NA | NA | NA
Epistaxis (Vascular disorders) | 63 | 43 | 0 | NA | NA | NA
Flushing (Vascular disorders) | 19 | 14 | 0 | NA | NA | NA
Hot flush (Vascular disorders) | 27 | 32 | 0 | NA | NA | NA
Hypertension (Vascular disorders) | 22 | 37 | 0 | NA | NA | NA
Lymphoedema (Vascular disorders) | 17 | 12 | 0 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.